CLINICAL TRIAL: NCT04730609
Title: Dexmedetomidine for Treatment of Shivering During Scheduled Elective Cesarean Delivery: Determining the Optimal Dose
Brief Title: Dexmedetomidine for Intraoperative Shivering in Scheduled Elective Cesarean Delivery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hans P. Sviggum, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-004712
Record Dates: First submitted 2021-01-18; First posted 2021-01-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Shivering; Dose Finding Study
Keywords: Shivering; Cesarean Delivery; Dexmedetomidine; Dosing
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dexmedetomidine (Experimental): IV administration of Dexmedetomidine, using an Up-Down method utilizing a biased coin design to determine that next patient's dose. Initial dose will be 10mcg.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Doses of dexmedetomidine will be selected according to a sequential up-and-down method, using a biased coin design to find the estimated dose at which 90% of patients would have desired effect

SUMMARY:
The purpose of this study is to determine the optimum dose of Dexmedetomidine to stop shivering in 90% of patients who experience shivering during scheduled elective cesarean deliveries.

DETAILED DESCRIPTION:
Potential subjects will consist of parturients who present for scheduled elective cesarean deliveries. Patients will be recruited and consented for the study pre-operatively and if they display Grade 3 or 4 shivering at the time of delivery then they will be enrolled in the study. Doses of dexmedetomidine will be selected according to a sequential up-and-down method, using a biased coin design to find the estimated dose at which 90% of patients would have desired effect - cessation of shivering within 5 minutes of medication administration. An anesthesia physician not involved in patient care or assessment will prepare the dexmedetomidine for intravenous use. Anesthesia will be initiated with spinal anesthesia with our institution's typical dosing of 1.6 mL 0.75% bupivacaine with dextrose, 15 mcg fentanyl, and 150 mcg morphine.

Shivering will be graded using a five-point scale as outlined by Crossley and Mahajan. Members of the anesthesia team caring for women in the study will be educated on the grading scales.

* Grade 0: no shivering;
* Grade 1: one or more of the following: piloerection, peripheral vasoconstriction, peripheral cyanosis, but without visible muscle activity; Grade 2: visible muscle activity confined to one muscle group;
* Grade 3: visible muscle activity in more than one muscle group;
* Grade 4: gross muscle activity involving the whole body

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for planned cesarean delivery.
* American Society of Anesthesiology Physical Classification Status 2 or 3; without major medical co-morbidities.
* Singleton gestation in the 3rd trimester (28-42 weeks gestation).
* Spinal anesthesia technique Women presenting for planned cesarean delivery.
* American Society of Anesthesiology Physical Classification Status 2 or 3; without major medical co-morbidities.
* Singleton gestation in the 3rd trimester (28-42 weeks gestation).
* Spinal anesthesia technique.

Exclusion Criteria:

* Any contraindication to spinal anesthesia technique.
* Allergy or intolerance to dexmedetomidine or clonidine.
* Oral temperature < 36° Celsius prior to procedure.
* Unable to give personal consent.
* PPROM or concern for infection (e.g., chorioamnionitis).
* Conversion to General Anesthesia prior to randomization.
* Sedative medications (e.g., fentanyl, midazolam, ketamine, nitrous oxide) administered prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Shivering will be graded using a five-point scale as outlined by Crossley and Mahajan | 5 minutes after administration of the drug
  Cessation of shivering

SECONDARY OUTCOMES:
Maternal Heart Rate | During intraoperative course
  Determination of the effect of varying doses of dexmedetomidine on maternal heart rate.
Doses of dexmedetomidine | During intraoperative course
  Determination of the effect of varying doses of dexmedetomidine on maternal sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Sviggum, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No